CLINICAL TRIAL: NCT05611749
Title: Postoperative Duloxetine Impact on Pain Control and Patient Outcomes Following Lateral Lumbar Interbody Fusion: A Randomized Controlled Trial
Brief Title: Duloxetine Impact on Postoperative Pain Control and Outcomes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment was extremely low and there were too many adverse events.
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, Gregory M. Mundis Jr., MD, Pediatric and Adult Spinal Deformity Surgery Co-Director San Diego Spine Fellowship Scripps Clinic Division of Orthopedic Surgery, Scripps Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-21-7830
Record Dates: First submitted 2022-08-02; First posted 2022-11-10 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Acute Post-operative Pain; Chronic Post Operative Pain; Narcotic Use; Opioid Use; Opioid Addiction
Keywords: Acute pain; Chronic pain; narcotic consumption; patient outcomes
MeSH Terms: conditions — Pain, Postoperative; Opioid-Related Disorders; Acute Pain; Chronic Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either a control group receiving a placebo (n=65) or a treatment group receiving 60 mg Duloxetine (a selective serotonin and norepinephrine reuptake inhibitor) (n=65). Surgeons, patients, research staff, PACU staff, and floor staff will be blinded to group allocation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized on the day of surgery in the preoperative area by the investigational pharmacist, who will be the only staff unblinded. The study medication (either placebo or Duloxetine) will be continued throughout the duration of hospitalization. The balance of the remaining pills will be provided to the patient as a discharge prescription to allow for 10 days total treatment via 'Meds to Beds.'
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- control group receiving a placebo (Placebo Comparator): The study medication (either placebo or Duloxetine) will be continued throughout the duration of hospitalization. The balance of the remaining pills will be provided to the patient as a discharge prescription to allow for 10 days total treatment.
  Interventions: Other: Placebo
- treatment group receiving 60 mg Duloxetine (Experimental): The study medication (either placebo or Duloxetine) will be continued throughout the duration of hospitalization. The balance of the remaining pills will be provided to the patient as a discharge prescription to allow for 10 days total treatment.
  Interventions: Drug: Duloxetine 60 MG

INTERVENTIONS:
Drug: Duloxetine 60 MG — Looking at the use of duloxetine's effect with regards to perioperative narcotics consumption and patient outcomes after lumbar fusion.
  Other Names: Drizalma Sprinkle; Cymbalta; Irenka
  Arms: treatment group receiving 60 mg Duloxetine
Other: Placebo — Duloxetine versus placebo in reducing postoperative narcotic consumption among patients undergoing lateral lumbar interbody fusions
  Arms: control group receiving a placebo

SUMMARY:
1. Evaluate differences between patients taking Duloxetine or placebo following lateral lumbar interbody fusion for postoperative narcotic consumption.
2. Evaluate differences between patients taking Duloxetine or placebo following lateral lumbar interbody fusion for postoperative pain, function, and quality of life.
3. Evaluate the correlation between preoperative screening tests (measuring pain centralization, anxiety, depression, and overall function) and patients' response to treatment (reduction in pain, anxiety, or depression and improvement in function).

DETAILED DESCRIPTION:
It is widely accepted that over-prescription of narcotics by medical providers has played a significant role in the recent uptick in the nationwide opioid crisis facing American society. As such, a tremendous amount of research within the surgical community has been dedicated to reducing the need for narcotics in the acute postoperative period. Anti-depressants, including tricyclics as well as selective serotonin inhibitors (both SSRIs and SNRIs), have been identified in several trials as having potential benefit for treating acute postoperative pain.

Duloxetine (an SNRI) has been approved by the FDA for treating mental health conditions such as depression and anxiety as well as chronic musculoskeletal pain. Previous studies have established its efficacy in treating acute postoperative pain following orthopaedic procedures such as total joint arthroplasty, even with relatively short durations of treatment. Specifically, previous randomized controlled trials have demonstrated that perioperative duloxetine leads to decreased narcotics consumption as well as improved function scores in patients undergoing total knee arthroplasty.

While there has been a fair amount of research within the arthroplasty literature, there is minimal research to date investigating the potential benefits of this medication in the spine literature. Lateral interbody fusion is a commonly performed procedure where an interbody spacer (typically made of either PEEK or titanium) is placed between two adjacent vertebrae. This is usually done with the goal of increasing the space between the bones and/or to fuse the two bones together, thereby reducing the amount of motion that occurs during activities of daily living. To this point, there has not been any studies looking at the use of duloxetine's effect with regards to perioperative narcotics consumption and patient outcomes after lumbar fusion.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 24 years
* Male / Female not meeting any of the exclusion criteria

Exclusion Criteria:

* Age < 24 years
* Current use of antidepressant medications (including SSRI/SNRI, tricyclic, or Monoamine Oxidase Inhibitors)
* History of seizure disorder
* Diagnosis of bipolar disorder
* History of syncope/orthostatic hypotension
* Diagnosis of any condition with slowed gastric emptying
* History of suicidal ideation
* History of liver disease
* History of chronic kidney disease/renal impairment
* History of angle-closure glaucoma.

Ages: 24 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Evaluating the amount of change in pain, for patients prescribed Duloxetine versus those patients prescribed the placebo following lateral lumbar interbody fusion | The study medication (either placebo or Duloxetine) will be continued throughout the duration of hospitalization. Remaining pills will be provided to the patient as a discharge prescription to allow for 10 days total treatment.
  Evaluate the effectiveness of Duloxetine versus placebo through the assessment of postoperative narcotic consumption.
Measuring the amount of change in pain, for patients prescribed Duloxetine versus those patients prescribed the placebo following lateral lumbar interbody fusion | The study medication (either placebo or Duloxetine) will be continued throughout the duration of hospitalization. Remaining pills will be provided to the patient as a discharge prescription to allow for 10 days total treatment.
  Measure the differences between patients taking Duloxetine or placebo following lateral lumbar interbody fusion for postoperative pain.
Evaluating the amount of change in function for patients prescribed Duloxetine versus those patients prescribed the placebo following lateral lumbar interbody fusion | The study medication (either placebo or Duloxetine) will be continued throughout the duration of hospitalization. Remaining pills will be provided to the patient as a discharge prescription to allow for 10 days total treatment.
  Evaluate the effectiveness of Duloxetine versus placebo through the assessment of postoperative narcotic consumption.
Measuring the amount of change in function for patients prescribed Duloxetine versus those patients prescribed the placebo following lateral lumbar interbody fusion | The study medication (either placebo or Duloxetine) will be continued throughout the duration of hospitalization. Remaining pills will be provided to the patient as a discharge prescription to allow for 10 days total treatment.
  Measure the differences between patients taking Duloxetine or placebo following lateral lumbar interbody fusion for postoperative pain.
Evaluating the amount of change in narcotic consumption for patients prescribed Duloxetine versus those patients prescribed the placebo following lateral lumbar interbody fusion | The study medication (either placebo or Duloxetine) will be continued throughout the duration of hospitalization. Remaining pills will be provided to the patient as a discharge prescription to allow for 10 days total treatment.
  Evaluate the effectiveness of Duloxetine versus placebo through the assessment of postoperative narcotic consumption.
Measuring the amount of change in narcotic consumption for patients prescribed Duloxetine versus those patients prescribed the placebo following lateral lumbar interbody fusion | The study medication (either placebo or Duloxetine) will be continued throughout the duration of hospitalization. Remaining pills will be provided to the patient as a discharge prescription to allow for 10 days total treatment.
  Measure the differences between patients taking Duloxetine or placebo following lateral lumbar interbody fusion for postoperative pain.
Measuring the general domains of health with PROMIS Global questionnaire | Patients will be asked to complete the PROMIS Global at baseline visit
  The PROMIS Global questionnaire is a patient reported outcome that evaluates and identifies the life domains in areas such as physical, mental and social health. Scoring for the questionnaire is out of 50 points and the higher the score the healthier the patient.
Measuring the general domains of function with PROMIS Global questionnaire | Patients will be asked to complete the PROMIS Global at baseline visit
  The PROMIS Global questionnaire is a patient reported outcome that evaluates and identifies the life domains in areas such as physical, mental and social health. Scoring for the questionnaire is out of 50 points and the higher the score the healthier the patient.
Measuring the general domains of health with PROMIS Global questionnaire | Patients will be asked to complete the PROMIS Global at 2 week post-op visit
  The PROMIS Global questionnaire is a patient reported outcome that evaluates and identifies the life domains in areas such as physical, mental and social health. Scoring for the questionnaire is out of 50 points and the higher the score the healthier the patient.
Measuring the general domains of function with PROMIS Global questionnaire | Patients will be asked to complete the PROMIS Global at 2 week post-op visit
  The PROMIS Global questionnaire is a patient reported outcome that evaluates and identifies the life domains in areas such as physical, mental and social health. Scoring for the questionnaire is out of 50 points and the higher the score the healthier the patient.
Measuring the general domains of health with PROMIS Global questionnaire | Patients will be asked to complete the PROMIS Global at 4 week post-op visit
  The PROMIS Global questionnaire is a patient reported outcome that evaluates and identifies the life domains in areas such as physical, mental and social health. Scoring for the questionnaire is out of 50 points and the higher the score the healthier the patient.
Measuring the general domains of function with PROMIS Global questionnaire | Patients will be asked to complete the PROMIS Global at 4 week post-op visit
  The PROMIS Global questionnaire is a patient reported outcome that evaluates and identifies the life domains in areas such as physical, mental and social health. Scoring for the questionnaire is out of 50 points and the higher the score the healthier the patient.
Measuring the general domains of health with PROMIS Global questionnaire | Patients will be asked to complete the PROMIS Global at 8 week post-op visit
  The PROMIS Global questionnaire is a patient reported outcome that evaluates and identifies the life domains in areas such as physical, mental and social health. Scoring for the questionnaire is out of 50 points and the higher the score the healthier the patient.
Measuring the general domains of function with PROMIS Global questionnaire | Patients will be asked to complete the PROMIS Global at 8 week post-op visit
  The PROMIS Global questionnaire is a patient reported outcome that evaluates and identifies the life domains in areas such as physical, mental and social health. Scoring for the questionnaire is out of 50 points and the higher the score the healthier the patient.
Patient's anxiety symptoms severity at baseline visit | Patients will be asked to complete the GAD-7 at the baseline visit
  The Generalized Anxiety Disorder-7 (GAD-7) is an assessment tool to measure the changes in a treatments progress and provide guidance for treatment decisions, interventional targets and give assistance in differential diagnosis. Scoring for this measure is based off the patient reporting anxiety symptoms on a Likert scale. The scale scoring is rom 1- 21. The lower the score the less the severity of anxiety symptoms being reported by a patient.
Patient's anxiety symptoms severity at eight week visit | Patients will be asked to complete the GAD-7 at the 8 week post-op visit.
  The Generalized Anxiety Disorder-7 (GAD-7) is an assessment tool to measure the changes in a treatments progress and provide guidance for treatment decisions, interventional targets and give assistance in differential diagnosis. Scoring for this measure is based off the patient reporting anxiety symptoms on a Likert scale. The scale scoring is rom 1- 21. The lower the score the less the severity of anxiety symptoms being reported by a patient.
Measuring a patient's baseline visit for severity of depression symptoms with Beck's Depression Inventory | Patient s will complete the Beck's Depression Inventory at the baseline visit.
  The Beck's Depression Inventory questionnaire is a patient self-reporting measurement of a patients symptoms and the related characteristic and attitudes pertaining to depression. This measure is cored on a scale 0-3 on 21 questions. The higher the score the worse the outcome is for the severity of depression.
Measuring a patient's eight week visit for severity of depression symptoms with Beck's Depression Inventory | Patient s will complete the Beck's Depression Inventory at the 8 week post-op visit.
  The Beck's Depression Inventory questionnaire is a patient self-reporting measurement of a patients symptoms and the related characteristic and attitudes pertaining to depression. This measure is cored on a scale 0-3 on 21 questions. The higher the score the worse the outcome is for the severity of depression.
Measuring at the baseline of a patient's hypersensitivity to noxious and non-noxious stimuli with the Central Sensitization Inventory | Patients will complete the Central Sensitization Inventory at the baseline visit.
  The Central Sensitization inventory is a patient self reporting on the severity of their central sensitization pain they are experiencing. The pain severity is scored from 0-100 ( (subclinical= 0-29), (mild=30-39), (moderate=40-49), (severe= 50-59) and (extreme=60-100). The higher the score equates to the worse the outcome.
Measuring at eight weeks to evaluate a patient's hypersensitivity to noxious and non-noxious stimuli with the Central Sensitization Inventory | Patients will complete the Central Sensitization Inventory at the 8 week post-op visit.
  The Central Sensitization inventory is a patient self reporting on the severity of their central sensitization pain they are experiencing. The pain severity is scored from 0-100 ( (subclinical= 0-29), (mild=30-39), (moderate=40-49), (severe= 50-59) and (extreme=60-100). The higher the score equates to the worse the outcome.
Baseline to measure a patient's catastrophic thinking in relation to adults with or without chronic pain. | The patient will complete the Pain Catastrophizing Scale at the baseline visit.
  The Pain Catastrophizing Scale is measure that a patient self-reports their thoughts and feelings that may be associated to the pain that they may or may not be experiencing. The scoring of this scale is as follows: 0=not at all, 1=to a slight degree, 2=to a moderate degree, 3= to a great degree, 4= all the time. The higher the score equals the worse the outcome
Eight week measurement of a patient's catastrophic thinking in relation to adults with or without chronic pain. | The patient will complete the Pain Catastrophizing Scale at the 8 week post-op visit.
  The Pain Catastrophizing Scale is measure that a patient self-reports their thoughts and feelings that may be associated to the pain that they may or may not be experiencing. The scoring of this scale is as follows: 0=not at all, 1=to a slight degree, 2=to a moderate degree, 3= to a great degree, 4= all the time. The higher the score equals the worse the outcome
Two week evaluation of amount of change in post-op pain improvement | Patients to be evaluated at post-op at 2 weeks.
  Evaluate the correlation between preoperative screening tests (measuring pain centralization, anxiety, depression, and overall function) and patients' response to treatment (reduction in pain, anxiety, or depression and improvement in function). Continued use of previously mentioned patient reported outcomes will be measured at the designated time points
Four week evaluation of amount of change in post-op pain improvement | Patients to be evaluated at post-op at 4 weeks.
  Evaluate the correlation between preoperative screening tests (measuring pain centralization, anxiety, depression, and overall function) and patients' response to treatment (reduction in pain, anxiety, or depression and improvement in function). Continued use of previously mentioned patient reported outcomes will be measured at the designated time points
Eight week evaluataion of amount of change in post-op pain improvement | Patients to be evaluated at post-op at 8 weeks.
  Evaluate the correlation between preoperative screening tests (measuring pain centralization, anxiety, depression, and overall function) and patients' response to treatment (reduction in pain, anxiety, or depression and improvement in function). Continued use of previously mentioned patient reported outcomes will be measured at the designated time points
Two week evaluation of amount of change in post-op quality of life improvement | Patients to be evaluated at post-op at 2 weeks
  Evaluate the correlation between preoperative screening tests (measuring pain centralization, anxiety, depression, and overall function) and patients' response to treatment (reduction in pain, anxiety, or depression and improvement in function). Continued use of previously mentioned patient reported outcomes will be measured at the designated time points
Four week evaluation of amount of change in post-op quality of life improvement | Patients to be evaluated at post-op at 4 weeks.
  Evaluate the correlation between preoperative screening tests (measuring pain centralization, anxiety, depression, and overall function) and patients' response to treatment (reduction in pain, anxiety, or depression and improvement in function). Continued use of previously mentioned patient reported outcomes will be measured at the designated time points
Eight week evaluation of amount of change in post-op quality of life improvement | Patients to be evaluated at post-op at 8 weeks.
  Evaluate the correlation between preoperative screening tests (measuring pain centralization, anxiety, depression, and overall function) and patients' response to treatment (reduction in pain, anxiety, or depression and improvement in function). Continued use of previously mentioned patient reported outcomes will be measured at the designated time points

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Mundis, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Clinic Torrey Pines, La Jolla, California, United States